CLINICAL TRIAL: NCT05894109
Title: Efficacy of Zinc Supplementation on Botox Treated Forehead Rhytids
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Per the PI, the project is not IRB approved yet and will likely not be completed.
Sponsor: University of New Mexico (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Jeffrey Wu, Associate Professor of Surgery, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00006041
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Adjuvant Zinc May Increase the Efficacy of Botulinum Toxin; Zinc Supplementation for Botulinum Toxin Treatment of the Forehead; Glabellar Frown Lines; Botulinum Toxin, Cosmetic; Adjuvant Oral Zinc and Botulinum Toxin

STUDY DESIGN:
Intervention Model Description: Repeated Measures ANOVA (Continuous Data) McNemar Test (Categorical Data)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OnabotulinumtoxinA without Zinc Supplementation (Placebo Comparator): Given placebo
  Interventions: Other: Placebo Microcrystalline Cellulose
- OnabotulinumtoxinA with Zinc Supplementation (Experimental): Given 50 mg of zinc citrate
  Interventions: Dietary Supplement: zinc citrate 50 mg

INTERVENTIONS:
Dietary Supplement: zinc citrate 50 mg — will take zinc citrate 4 days before and 1 week after botulinum toxin injection
  Arms: OnabotulinumtoxinA with Zinc Supplementation
Other: Placebo Microcrystalline Cellulose — will take placebo 4 days before and 1 week after botulinum toxin injection
  Other Names: Capsulated Microcrystalline Cellulose
  Arms: OnabotulinumtoxinA without Zinc Supplementation

SUMMARY:
The current literature suggests that zinc supplementation may increase the duration of botulinum toxin; however, each study had their limitations. Further, no one has studied the effect of zinc supplementation for botulinum toxin treatment of the forehead. The purpose of this study is to evaluate the effect of zinc supplementation on frontalis muscle denervation by objectively assessing the degree of forehead rhytids and movement of the eyebrows.

ELIGIBILITY:
Inclusion Criteria:

Any patient older than 18 years old who desires botulinum toxin injection to decrease forehead rhytids

Exclusion Criteria:

* Allergy to any components of zinc citrate or botulinum toxin
* inflammation or infection at site of injection
* patients using anticholineresterase or other agents interfering with neuromuscular transmission
* patients with any medical condition that can affect frontalis function (Bell's palsy, Möbius syndrome, Hemifacial microsomia, CHARGE syndrome, stroke, etc)
* patients with any prior trauma that could have potentially injured the frontalis muscle
* patients dependent on intact facial movements and expressions for their livelihood (actors, singers, musicians, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Duration of botulinum toxin on eyebrow excursion | 1 year
  Measurement of eyebrow excursion
Duration of botulinum toxin effect on forehead rhytids | 1 year
  Visual assessment of return of forehead rhytids

SECONDARY OUTCOMES:
Side effects of zinc administration | 1 year
  Monitor for adverse side effects of adjunct oral zinc therapy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koshy JC, Sharabi SE, Feldman EM, Hollier LH Jr, Patrinely JR, Soparkar CN. Effect of dietary zinc and phytase supplementation on botulinum toxin treatments. J Drugs Dermatol. 2012 Apr;11(4):507-12. PMID 22453589
- [Result] Shemais N, Elarab AE, ElNahass H. The effect of botulinum toxin A in patients with excessive gingival display with and without zinc supplementation: randomized clinical trial. Clin Oral Investig. 2021 Nov;25(11):6403-6417. doi: 10.1007/s00784-021-03944-2. Epub 2021 May 5. PMID 33950373